CLINICAL TRIAL: NCT04215640
Title: Radiofrequency Ablation of Paroxysmal Supraventricular Tachycardia Using a Novel Catheter Equipped With Mini Electrodes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yong Seog Oh (Other)
Responsible Party: Sponsor-Investigator, Yong Seog Oh, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XC19DEDI0078K
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Paroxysmal Supraventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Catheters

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIFI group (Experimental): Patients in the MIFI group receive standard radiofrequency ablation procedure for the supraventricular tachycardia using microfidelity (MIFI) catheter.
  Interventions: Device: Microfidelity (MIFI) catheter
- Control (Active Comparator): Patients in the control group receive standard radiofrequency ablation procedure for the supraventricular tachycardia using conventional ablation catheter (Blazer II).
  Interventions: Device: Conventional ablation catheter

INTERVENTIONS:
Device: Microfidelity (MIFI) catheter — Patients are randomized into the MIFI group and control group. Radiofrequency ablation will target slow pathway for AVNRT or accessory pathway for AVRT. Microfidelity (MIFI) catheter equipped with mini-electrodes will be used for ablation in the MIFI group.
  Arms: MIFI group
Device: Conventional ablation catheter — Patients are randomized into the MIFI group and control group. Radiofrequency ablation will target slow pathway for AVNRT or accessory pathway for AVRT. Blazer II radiofrequency ablation catheter will be used for ablation in the control group.
  Arms: Control

SUMMARY:
Paroxysmal supraventricular tachycardia is treated with radiofrequency ablation recently. This procedure is performed by ablating slow pathway or accessory pathway using radiofrequency ablation catheter. Recently developed mirofidelity (MIFI) catheter has mini-electrodes that can record local eletrogram with higher resolution. We aimed to investigate the efficacy of MIFI catheter in the ablation of paroxysmal supraventricular tachycardia compared to conventional radiofrequency ablation catheter. Enrolled patients undergo conventional electrophysiologic study. Patients with sustained supraventricular tachycardia during the study are randomized to either study group or control group. Radiofrequency ablation is performed using MIFI catheter in the study group, and conventional catheter (Blazer II) in the control group. The study endpoints are recorded immediately after ablation and there is no additional follow up or management after procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo radiofrequency ablation for paroxysmal supraventricular tachycardia or WPW syndrome with atrial fibrillation
* Give written informed consent for the study

Exclusion Criteria:

* Unable to induce supraventricular tachycardia during electrophysiologic study.
* Cognitive impairment to understand study procedure

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
RF time (seconds) to successful ablation | At the end of radiofrequency ablation procedure
  For AVNRT, the time (seconds) from the beginning of radiofrequency ablation to the emergence of junctional rhythm For AVRT, the time (seconds) from the beginning of radiofrequency ablation to the accessory pathway block
RF application number | At the end of radiofrequency ablation procedure
  Number of radiofrequency ablation attempt to successful ablation

SECONDARY OUTCOMES:
Total ablation time (seconds) | At the end of radiofrequency ablation procedure
  Total time of radiofrequency energy delivery
Presence of either acute reconnection or reinduction | At the end of radiofrequency ablation procedure
  Acute accessory pathway reconnection or supraventricular tachycardia reinduction after ablation

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Seog Oh, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St Mary's Hospital, Seoul, Seo Ch-gu, South Korea

IPD SHARING:
Plan to Share IPD: No
IPD would be provided with an appropriate request from other investigators.

REFERENCES:
- [Derived] Choi Y, Kim SH, Kim H, Park JW, Ha YW, Hwang Y, Kim JH, Jang SW, Oh YS. The advantage of the mini-electrode-equipped catheter for the radiofrequency ablation of paroxysmal supraventricular tachycardia. J Cardiovasc Electrophysiol. 2022 Oct;33(10):2164-2171. doi: 10.1111/jce.15639. Epub 2022 Aug 24. PMID 35924472